CLINICAL TRIAL: NCT00435604
Title: Phase I Dose-Ranging Randomized Double-Blinded Controlled Study of the Subcutaneous Injection of a Viscous Antibody Solution With Recombinant Human Hyaluronidase
Brief Title: A Study of the Subcutaneous Injection of a Viscous Antibody Solution With Recombinant Human Hyaluronidase
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Halozyme Therapeutics (Industry)
Responsible Party: Richard Yocum, M.D., Vice President of Clinical Dev and Med Affairs, Halozyme Therapeutics
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: HZ2-07-01
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2007-02

CONDITIONS: Healthy
Keywords: hyaluronidase; subcutaneous drug delivery; Volunteer Subjects

INTERVENTIONS:
Drug: Hylenex

SUMMARY:
This Phase I, randomized, double-blinded, within-subject controlled, two-way crossover study comparing the time to inject (flow rate), safety, and tolerability of a subcutaneously (SC) administered, viscous antibody solution of with and without human recombinant hyaluronidase (rHuPH20) in volunteer subjects.

The study hypothesizes that the time required to complete a 20-mL SC injection of a viscous antibody with rHuPH20 will be comparable or shorter than the time required for the injection without rHuPH20.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers of either sex, age 18 to 65 years, inclusive.
2. Intact normal skin on both upper extremities without tattoos or potentially obscuring pigmentation or lesions.
3. Vital signs (BP, HR, temperature, respiratory rate) within normal range.
4. Metabolic panel (e.g., sodium, potassium, chloride, bicarbonate, BUN, creatinine, glucose, calcium, AST, ALT, alkaline phosphatase, total bilirubin, albumin, and total protein) within normal range within 7 days of injection.
5. A negative serum or urine pregnancy test (if female of child-bearing potential) within 7 days of injection.
6. Female subjects of child-bearing potential must be practicing effective birth control or abstinence currently and plan to continue to do so for the duration of the study.
7. Decision-making capacity and willingness and ability to comply with the requirements for full completion of the trial.
8. Willingness and ability to sign an informed consent document.

Exclusion Criteria:

1. Upper extremity edema.
2. Upper extremity pathology that could interfere with any protocol-specified outcome assessment (e.g., cellulitis, lymphatic disorder or prior surgery, preexisting pain syndrome, previous mastectomy and/or axillary lymph node dissection, etc.).
3. Contraindication to an antibody, such as known history of anaphylactic or severe systemic reactions.
4. Known predisposition to renal insufficiency or renal failure, including diabetes mellitus, volume depletion, sepsis, paraproteinemia, and subjects receiving known nephrotoxic drugs.
5. Known allergy to hyaluronidase or any other ingredient in the formulation of Hylenex.
6. Known allergy to bee or vespid venom.
7. Known coagulopathy.
8. Pregnancy or breast-feeding woman.
9. Known clinically significant cardiovascular, gastrointestinal, hepatic, neurological, psychiatric, endocrine, cancer, HIV infection, diabetes mellitus, intercurrent illness such as influenza, or other major systemic disease that would unduly risk the subject's safety or interfere with the interpretation of results.
10. Participation in a study of any investigational drug or device within 30 days of enrollment in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2007-02; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
The time to inject 20 mL of a viscous antibody solution with and without rHuPH20.

SECONDARY OUTCOMES:
Assess the time required for a subcutaneous injection with various doses of rHuPH20, safety, tolerability.

CONTACTS AND LOCATIONS:
Overall Officials: Anoshie Ratnayake, M.D., Principal Investigator — Principal Investigator